CLINICAL TRIAL: NCT06779188
Title: Treating Balance Impairment of the Elderly With TMS-induced Brain Connectivity
Brief Title: Examining the Effects of Theta Burst TMS on Brain Connectivity and Balance Ability in Older Adults With Balance Problems
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Weinberg Medical Physics LLC (Industry)
Collaborators: University of Houston (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004556; R41AG085838 (NIH)
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Aging; Balance Deficits
Keywords: TMS; Balance; Brain stimulation; Elderly; Treatment
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and their caregivers will not know whether they are receiving TMS or sham. The outcome assessors will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants in this group will receive transcranial magnetic stimulation (TMS) once daily, 5 days a week. TMS will be in the form of accelerated repetitive TMS. TMS is a safe technique when handled by experts.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham group (Sham Comparator): Participants in this group will receive sham (placebo) TMS once daily, 5 days a week.
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS (in the form of theta burst stimulations) will be delivered over Supplementary Motor Area while the subject is seated in the Treatment group. TMS is capable to induce neuroplastic facilitatory changes in the brain that last beyond the duration of stimulation. TMS will be delivered once daily, 5 days per week, for 4 weeks.
  Arms: Treatment group
Device: Transcranial Magnetic Stimulation Sham — Sham TMS will be delivered in the sham group using a sham coil once daily, 5 days per week, for 4 weeks.
  Arms: Sham group

SUMMARY:
The goal of this study is to learn if manipulating the brain using magnets works to treat balance impairment, a major cause of falls, in older adults with balance problems. The technique to manipulate the brain using magnets is known as transcranial magnetic stimulation or TMS.

The main questions this study aims to answer are:

* How does TMS change communication between brain areas?
* Does TMS improve balance ability in older adults with balance problems? Researchers will compare the TMS group to a placebo group to see if manipulating the brain using magnets works to treat balance impairment.

Participants will:

* Receive TMS or placebo stimulation for 4 weeks.
* Visit the laboratory for checkups and tests 3 times.

DETAILED DESCRIPTION:
Falls and fall-related injuries are a growing public health concern, particularly in regions of the world in which high proportions of the population are elderly. When these older adults are affected with neurological conditions such as stroke, neuropathies, Parkinson's disease, Alzheimer's disease, the risk for falls increases more than 3-fold. Falls and the resulting fear of falls can mark the beginning of a decline in function, participation in social activities, and independence, thus negatively affecting the quality of life.

The aim of this project is to use electroencephalography-guided TMS to improve balance in elderly patients with a history of falls, through repair of (or compensation for) abnormal brain connectivity. The entire study will be done at the University of Houston in Dr. Parikh's laboratory (PI) in the Center for Neuromotor and Biomechanics laboratory (CNBR).

The investigators will enroll 30 older adults with balance problems. Participants will be randomly and equally assigned to a treatment group (A) and a placebo (sham) group (B). Each participant will undergo a MRI scan at the MRI center. Participants will not be responsible for MRI-related costs. This will be followed by baseline assessments of brain connectivity using electroencephalography (EEG) and balance assessment. Participants in both groups will receive a 4-week long intervention (once daily, 5 days a week). Immediately following the intervention period, EEG and balance assessments will be repeated. A 3-month follow-up will be conducted.

ELIGIBILITY:
Inclusion Criteria:

a) Able to provide informed consent b) All ethnic groups c) >65 years of age d) ≥2 non-injury falls or ≥1 injury fall in the past year [17]-[21] e) Absence of dementia/uncontrolled psychiatric disorder h) Able to walk and stand for 5 min continuously independently without assistance (i.e., cane, walker, ankle foot orthotics, electric scooter).

i) Willingness to undergo MRI, participate in the 4-weeks intervention AND in the laboratory studies before, immediately-after, and 3-month after the intervention.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Non-English speaking.
3. Have contraindications to TMS based on TMS Adult Safety Screen (e.g., pregnancy, metal in the brain/skull, neurostimulator, pacemaker, infusion device, medication to treat mental illness)
4. Unintentional weight loss of ≥10 pounds over the past year.
5. Severe uncontrolled hypertension, or uncontrolled diabetes.
6. Poor cognitive status (Montreal Cognitive Assessment (MoCA) score ≥ 26)
7. Untreated depression or Geriatric Depression Scale score on 15 item scale >7
8. History of limb amputation (upper or lower extremity)
9. Planned surgery in the next 3 months.
10. History of chemotherapy or planned chemotherapy in the next 6 months or active malignancy.
11. Severe osteoporosis, defined by diagnosis of osteoporosis with fracture.
12. Pregnant or have a chance of being pregnant.
13. Chronic inflammatory condition, autoimmune disease or infectious processes such as active tuberculosis, Human Immunodeficiency Virus, Rheumatoid arthritis, systemic lupus erythematosus, acute or chronic hepatitis B or C.
14. Illicit drug use
15. Use of medications that may increase the risk of falling:

    * Sedatives
    * Hypnotics
    * Anti-cholinergic
    * Benzodiazepines
    * Anti-depressants
16. Intracranial bleeds visible on their most recent CT or MRI scans.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography functional connectivity | Before and immediately-after the intervention and at 3- month follow-up
  Electroencephalography (EEG) will be used to measure the brain activity. The brain circuitry responsible for balance will be evaluated with EEG projected onto individual anatomical MRI. Directed functional connectivity between two regions of activation will be computed. The higher the functional connectivity coefficient, the stronger the connectivity.
miniBESTest | Before and immediately-after the intervention and at 3- month follow-up
  It provides a comprehensive assessment of anticipatory and reactive postural control, sensory orientation, and dynamic gait.

SECONDARY OUTCOMES:
Activities-Specific Balance Confidence scale (Aim 2) | Before and immediately-after the intervention and at 3- month follow-up
  It consists of 16 items describing different situations that might lead to a loss of balance. For each time, scoring is done from 0-100 (0 is no confidence and 100 is full confidence). The total score is calculated by adding up all the individual item scores and dividing by 16. The Activities-Specific Balance Confidence total score is known to predict falls in elderly subjects.
Root mean square of foot center of pressure on the balance task | Before and immediately-after the intervention and at 3- month follow-up
  It is calculated from the ground reaction forces.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Neuromotor and Biomechanics Research at the University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided